CLINICAL TRIAL: NCT00154856
Title: Influence of Mechanical Stimulus on Distraction Osteogenesis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 92002015
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2005-09-12 (Estimated); Status verified 2003-02

CONDITIONS: Leg Discrepancy
Keywords: osteogenesis; Ilizarov fixator; motion analysis; FEM; bone stress

INTERVENTIONS:
Behavioral: Detect the variation of limb lengthening

SUMMARY:
a further step of our current one-year NSC project, aiming to bridge the above-mentioned gap by continuously monitoring the mechanical stimuli applied to the limb and callus, both through experimental measurements and FEM calculations, and by correlating the observed quantity and quality of the mechanical stimuli with the calculated stress and strain patterns of the callus tissue.

DETAILED DESCRIPTION:
Bone lengthening using distraction osteogenesis has found many clinical applications in the treatment of limb length discrepancies, limb deformities, bone defects and fracture nonunion. Animal studies have shown that mechanical conditions significantly affect the biological process of osteogenesis. Knowledge of the influence of mechanical stimuli on the formation of bone is thus essential for the improvement of the current technique, contributing to the treatment and care of patients receiving bone lengthening. Previous in vivo human studies have approached the problem by measuring the interfragmentary movement of bone fracture and the loading in the limb in terms of the ground reaction forces. The mechanical environment in the callus is not available with these approaches. As the stress and strain behavior of bone is critical to its normal function, the response to bone osteotomy and osteogenesis, a limited number of studies have used simplified FEM technique to examine the strain and stress patterns in the callus in two dimensions during simplified loading conditions. The calculated strain patterns, however, can be far from the real situation in the callus. No data are available for the stress and strain patterns during the process of distraction osteogenesis.

The present study is a further step of our current one-year NSC project, aiming to bridge the above-mentioned gap by continuously monitoring the mechanical stimuli applied to the limb and callus, both through experimental measurements and FEM calculations, and by correlating the observed quantity and quality of the mechanical stimuli with the calculated stress and strain patterns of the callus tissue. Specifically, in this proposed study, 3D finite element models of the osteogenesis at four temporal points during the limb lengthening process for each subject will be developed from CT data of the osteotomy sites. A 3D model of the musculoskeletal model of the lower limb will be used to calculate the forces transmitted by the bone and surrounding tissues, which will be used for subsequent FEM analysis. The purpose of the study is to determine the stress and strain patterns in the callus at different distraction stages and, with the data collected from gait laboratory experiments performed in our current NSC project, to provide a clearer picture of the influence of mechanical stimuli on distraction osteogenesis.

It is hoped that the present study will lead to a better understanding of the mechanisms of osteogenesis, which will be helpful in finding appropriate fixation methods in distraction osteogenesis that optimize the mechanical environment for bone formation.

ELIGIBILITY:
Inclusion Criteria:

* Leg differences above 3cm

Exclusion Criteria:

-

Min Age: 0 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10
Dates: Start 2004-08; Study Completion 2005-07

PRIMARY OUTCOMES:
Leg Length

CONTACTS AND LOCATIONS:
Overall Officials: Shier-Chieg Huang, MD, Study Chair — Dept. of Orthopaedic National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan